CLINICAL TRIAL: NCT01456832
Title: Post Operative Hyponatremia in the Renal Transplant Population
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, C. Burcin Taner, MD, Assistant Professor of Surgery, College of Medicine, Mayo Clinic
Other Study IDs: 11-004030
Record Dates: First submitted 2011-10-10; First posted 2011-10-21 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Hyponatremia
Keywords: hyponatremia; renal transplant
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal Transplant Patients with Post-operative Hypoatremia: All renal transplant recipients at the Mayo Clinic of Florida from 1/1/2010 through 8/19/2011 who received a kidney from either a living or cadaveric donor.

SUMMARY:
This study is designed to determine the causes of low sodium (salt) in the body fluids outside the cells for patients who have received a kidney transplant at the Mayo Clinic of Florida. The investigators will look at data collected on previous transplant patients at the Mayo Clinic to determine if the low sodium levels could be related to factors occurring in the course of surgery. The investigators hypothesize that the intravenous fluid used in the surgery, which is about half the concentration of normal saline, could contribute to the low sodium levels.

DETAILED DESCRIPTION:
This study is designed to determine the cause of post operative hyponatremia in renal transplant patients at the Mayo Clinic of Florida. Recently, the investigators have noted a trend in post-operative hyponatremia (low serum sodium) in patients who are recipients of both living donor and cadaveric kidneys. To improve the quality of care of this patient population, the investigators propose the investigation of the sources of this decline in serum sodium levels to determine if this is preventable. The investigators propose that a potential source of post-operative hyponatremia may be related to intra-operative factors. Currently, the intravenous fluid of choice used intra-operatively is 0.45% normal saline. The investigators hypothesize that this fluid choice contributes to post-operative hyponatremia.

To further investigate this the investigators will perform a retrospective review using the renal transplant database to collect data regarding pre-operative diagnoses, co-morbidities, and method of dialysis used in the pre-transplant period. Pre-operative serum sodium level will be compared to post-operative serum sodium levels. Data including post-operative complications, need and reasons for post-operative dialysis, and hospital course will also be collected. Once the data are analyzed and a primary source or sources are identified as causative agents for post-operative hyponatremia, an intervention to prevent a decline in serum sodium post-operatively will be planned for future study.

ELIGIBILITY:
Inclusion Criteria:

-Presenting to hospital for renal transplantation

Exclusion Criteria:

-Renal transplant recipients who received simultaneous transplantation of a liver, heart, or lung

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All renal transplant recipients who received a kidney transplant from either a living or cadaveric donor from 1/1/2010 through 8/19/2011 and subsequently developed post-operative hyponatremia.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2010-01; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Post-operative Hyponatremia Safety Issue?: Yes Incidence of Post-op Hyponatremia | up to 18 months
  To study the incidence of post operative hyponatremia in patients undergoing renal transplant at our institution.

SECONDARY OUTCOMES:
Etiology of hyponatremia | up to 18 months
  To evaluate potential causes of post operative hyponatremia in the renal transplant population at our institution.

CONTACTS AND LOCATIONS:
Overall Officials: Cemal Taner, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States